CLINICAL TRIAL: NCT00977236
Title: High Myopia - Partial Reduction Orthokeratology Study
Brief Title: Myopic Control for High Myopes Using Orthokeratology
Acronym: HM-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Procornea Nederland B.V. (Unknown)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-RP3M
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Myopia
Keywords: children; corneal reshaping; myopia; myopia control; orthokeratology
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orthokeratology lenses (Experimental): Children wearing orthokeratology at night for partial correction and spectacles at daytime for residual refractive error will be study group
  Interventions: Device: Orthokeratology lenses
- Single-vision spectacle lenses (Other): Children wearing single-vision spectacles in the daytime for correcting the refractive error will serve as control group
  Interventions: Device: Single-vision spectacle lenses

INTERVENTIONS:
Device: Orthokeratology lenses — Nightly use of orthokeratology to correct the refractive error and over-specs for a period of two years
  Other Names: Corneal reshaping therapy
  Arms: Orthokeratology lenses
Device: Single-vision spectacle lenses — Daily use of spectacles to correct the refractive error for a period of two years
  Other Names: Glasses; Spectacles
  Arms: Single-vision spectacle lenses

SUMMARY:
The purpose of this study is to evaluate and compare the eyeball elongation in high myopic children using partial correction orthokeratology and single-vision spectacles.

DETAILED DESCRIPTION:
Orthokeratology (ortho-k) has been shown to have strong potential for retardation of myopic progression in low myopes. To date, clinical experience has shown the technique to be less effective in achieving full myopic reduction in high myopes. Would myopic control be possible for high myopes undergoing partial correction ortho-k treatment?

A randomized, longitudinal study is designed to investigate the efficacy of partial correction ortho-k in retardation of myopic progression in high myopic children. Eye growth in terms of axial length elongation in children wearing ortho-k and over-spectacles (to correct residual refractive errors) (study group) and those wearing single-vision spectacles (control group) will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Myopia (refractive sphere): > 5.75D
* Astigmatism: < ½ of myopia; with-the-rule astigmatism (axes 180 +/- 30) ≤1.25D; astigmatism of other axes ≤ 0.50D
* Spherical equivalent (SE): > 5.75D
* Anisometropia: ≤ 1.50D in both refractive sphere, refractive cylinder and SE
* Best corrected monocular visual acuity: equal to or better than 0.10 in logMAR scale in both eyes
* Willingness for randomization
* Availability for follow-up for at least 2 years

Exclusion Criteria:

* Strabismus at distance or near
* Contraindication for contact lens wear and orthokeratology (e.g. limbus to limbus corneal cylinder and dislocated corneal apex
* Systemic or ocular conditions which may affect contact lens wear (e.g. allergy and medication)
* Systemic or ocular conditions which may affect refractive development (e.g. Down syndrome, ptosis)

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Determine the change in cycloplegic axial length in the study and control groups | 2 years

SECONDARY OUTCOMES:
Determine the incidence of adverse effects in cornea, the palpebral, bulbar and tarsal conjunctiva in the study and the control groups | 2 years
Rate of regression during the daytime | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Hong Kong SAR, China

REFERENCES:
- [Result] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Result] Walline JJ, Jones LA, Sinnott LT. Corneal reshaping and myopia progression. Br J Ophthalmol. 2009 Sep;93(9):1181-5. doi: 10.1136/bjo.2008.151365. Epub 2009 May 4. PMID 19416935
- [Result] Charm J, Cho P. High myopia-partial reduction ortho-k: a 2-year randomized study. Optom Vis Sci. 2013 Jun;90(6):530-9. doi: 10.1097/OPX.0b013e318293657d. PMID 23645372
- [Result] Charm J, Cho P. High myopia-partial reduction orthokeratology (HM-PRO): study design. Cont Lens Anterior Eye. 2013 Aug;36(4):164-70. doi: 10.1016/j.clae.2013.02.012. Epub 2013 Mar 18. PMID 23518209
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- See also: High myopia-partial reduction ortho-k: a 2-year randomized study — http://www.ncbi.nlm.nih.gov/pubmed/23645372
- See also: High myopia-partial reduction orthokeratology (HM-PRO): Study design. — http://www.ncbi.nlm.nih.gov/pubmed/23518209